CLINICAL TRIAL: NCT01087034
Title: Bracing During Infantile Scoliosis: Airways Study by Acoustic Method, EOS™ Acquisition and Noninvasive Respiratory Muscles Assessment
Brief Title: Bracing During Infantile Scoliosis: Airways Study
Acronym: MASI
Status: Completed | Type: Observational
Sponsor: Club d'Anesthésie-Réanimation Pédiatrique Armand Trousseau (Other)
Collaborators: Ecole Nationale Supérieure des Arts et Metiers (Unknown)
Responsible Party: Principal Investigator, Dr Nicolas LEBOULANGER, Dr, Club d'Anesthésie-Réanimation Pédiatrique Armand Trousseau
Other Study IDs: MA-SInf
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Scoliosis
Keywords: Infantile scoliosis; bracing; acoustic reflection method; EOS™; noninvasive; upper airways; thoracic penetration index; Idiopathic juvenile evolutive thoracic scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Milwaukee brace: Children with an infantile scoliosis requiring Milwaukee bracing
  Interventions: Device: Acoustic reflection method evaluation; Radiation: EOS™; Other: Non invasive respiratory muscle assessment
- Cheneaux brace: Children with an infantile scoliosis requiring Cheaneaux bracing
  Interventions: Device: Acoustic reflection method evaluation; Radiation: EOS™; Other: Non invasive respiratory muscle assessment

INTERVENTIONS:
Device: Acoustic reflection method evaluation — Evaluation of airways by acoustic relection method, with and without the bracing device
Radiation: EOS™ — Scoliosis and thoracic penetration index evaluation by EOS™ acquisition, with and without the bracing device
Other: Non invasive respiratory muscle assessment — Non invasive respiratory muscles assessment, with and without the bracing device.

SUMMARY:
Idiopathic juvenile thoracic scoliosis is a tridimensional deformation of the spine which may impact on the intrathoracic organs. Bracing is one of the oldest treatments of spinal deformities. It relies on the indirect manipulation of spinal curvatures in order to prevent curve progression, which may affect respiratory function.

The acoustic reflection method is based on the analysis of the reflection of a single transient planar wave giving the longitudinal cross-sectional area profile of the examined cavity. It is noninvasive and harmless.

The EOS™ device allows a double incidence, full body, and low-dose X-ray acquisition with thoracic 3D reconstruction.

The aim of the study is to evaluate the impact of bracing on the upper airways patency (by means of the acoustic method), on the breathing pattern (noninvasive respiratory muscles assessment), and on the thoracic penetration index (by means of the EOS™)

ELIGIBILITY:
Inclusion Criteria:

* children with evolutive juvenile thoracic scoliosis
* with a Cobb angle ≥ 30°
* requiring either a Milwaukee or a Cheneaux brace
* in a stable respiratory state

Exclusion Criteria:

* history of spine surgery

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with evolutive juvenile thoracic scoliosis requiring either a Milwaukee or a Cheneaux brace
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Impact of bracing on airways | 6 months
  The aim of the study is to evaluate the impact of bracing on the upper airways patency (by means of the acoustic method), on the breathing pattern (noninvasive respiratory muscles assessment), and on the thoracic penetration index (by means of the EOS™ system)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas LEBOULANGER, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Brigitte FAUROUX, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Armand Trousseau University Hospital, Paris
  - Ecole Nationale Supérieure des Arts et Metiers, Paris

REFERENCES:
- [Background] Donnelly LF, Bisset GS 3rd. Airway compression in children with abnormal thoracic configuration. Radiology. 1998 Feb;206(2):323-6. doi: 10.1148/radiology.206.2.9457181.
- [Background] Dubousset J, Charpak G, Skalli W, de Guise J, Kalifa G, Wicart P. [Skeletal and spinal imaging with EOS system]. Arch Pediatr. 2008 Jun;15(5):665-6. doi: 10.1016/S0929-693X(08)71868-2. No abstract available. French. PMID 18582707
- [Background] Heary RF, Bono CM, Kumar S. Bracing for scoliosis. Neurosurgery. 2008 Sep;63(3 Suppl):125-30. doi: 10.1227/01.NEU.0000320387.93907.97. PMID 18812914
- [Background] Jones RS, Kennedy JD, Hasham F, Owen R, Taylor JF. Mechanical inefficiency of the thoracic cage in scoliosis. Thorax. 1981 Jun;36(6):456-61. doi: 10.1136/thx.36.6.456. PMID 7314016
- [Background] Margonato V, Fronte F, Rainero G, Merati G, Veicsteinas A. Effects of short term cast wearing on respiratory and cardiac responses to submaximal and maximal exercise in adolescents with idiopathic scoliosis. Eura Medicophys. 2005 Jun;41(2):135-40. PMID 16200029